CLINICAL TRIAL: NCT00002804
Title: Phase II Study of Neoadjuvant Vincristine, Ifosfamide, Doxorubicin, and AND G-CSF in Children With Advanced Stage Non-Rhabdomyosarcoma Soft Tissue Sarcomas
Brief Title: Combination Chemotherapy, Surgery, and Radiation Therapy in Treating Children With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9553; POG-9553 (Other: Pediatric Oncology Group); CDR0000064905 (Other: Clinical Trials.gov); COG-P9953 (Other: Children's Oncology Group)
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Sarcoma
Keywords: nonmetastatic childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Doxorubicin; Ifosfamide; Mesna; Vincristine; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy Regimen (Experimental): Induction (Weeks 1-6) Vincristine sulfate (1.5 mg/m2) day 1, Ifosfamide (3 grams/m2) days 1-3, Doxorubicin (30 mg/m2) days 1-2, filgrastim day 4. Weeks 2 and 3 - Vincristine sulfate (1.5 mg/m2) IV day 1, week 5 no chemotherapy. Evaluate for response. Local Control (Weeks 7-13) Conventional surgery and radiation therapy. Vincristine sulfate (1.5 mg/m2) IV day 1, Ifosfamide (3 grams/m2) days 1-3, Doxorubicin (30 mg/m2) days 1-2, filgrastim day 4. Treatment continues per protocol.
  Interventions: Biological: filgrastim; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mesna; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: brachytherapy; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte-Colony Stimulating Factor; Neupogen; G-CSF
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC#123127
Drug: ifosfamide
  Other Names: Isophosphamide; IFEX
Drug: mesna
  Other Names: Sodium 2-Mercaptoethane Sulfonate; Mesnex; Urimetexan; NSC#113891
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC#67574
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, surgery, and radiation therapy in treating children who have advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response to vincristine/ifosfamide/doxorubicin (VID) with granulocyte colony-stimulating factor support in children with newly diagnosed, inoperable or metastatic non-rhabdomyosarcoma soft tissue sarcomas. II. Estimate the 2-year and event-free survival rates in children treated with VID plus radiotherapy and/or surgery. III. Establish a bank of frozen tumor and peripheral blood tissue for use in further molecular studies.

OUTLINE: The following acronyms are used: DOX Doxorubicin, NSC-123127 G-CSF Granulocyte Colony-Stimulating Factor (Amgen), NSC-614629 IFF Ifosfamide, NSC-109724 Mesna Mercaptoethane sulfonate, NSC-113891 VCR Vincristine, NSC-67574 VID VCR/IFF/DOX Induction: 3-Drug Combination Chemotherapy. VID. Local Control: Surgery and/or Radiotherapy plus 3-Drug Combination Chemotherapy. Excision of the primary tumor and pulmonary metastases; and/or irradiation of the primary tumor and pulmonary metastases using x-rays or Co60 beam energies of at least 4 MV (electrons or iridium-192 implant allowed for boost); plus VID. Continuation: 3-Drug Combination Chemotherapy. VID.

PROJECTED ACCRUAL: A total of 40 patients will be entered over 2.7 years if there are at least 7 responses in the first 20 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy proven non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) Evaluable residual tumor after initial biopsy or excision required Registration required within 42 days of definitive diagnosis Grade II/III, unresectable or metastatic disease The following histologies exclude: Angiofibroma of the nasopharynx Mesothelioma Desmoid tumor Peripheral neuroepithelioma Desmoplastic small cell tumor Rhabdomyosarcoma Extraosseous Ewing's sarcoma Undifferentiated sarcoma Kaposi's sarcoma Grade 1 NRSTS, including: Angiomatoid malignant fibrous histiocytoma Dermatofibrosarcoma protuberans Myxoid and well-differentiated liposarcoma Well-differentiated and infantile hemangiopericytoma Well-differentiated malignant peripheral nerve sheath tumor

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine normal for age No hydronephrosis Cardiovascular: Shortening fraction greater than 28% Other: No HIV infection Not pregnant or nursing Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy No prior nephrectomy (surgical correction of hydronephrosis allowed)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 1996-09; Primary Completion 2000-06 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Estimate the response rate to the combination of vincristine, ifosfamide, and doxorubicin (VID), with G-CSF support
  To estimate the response rate to the combination of vincristine, ifosfamide, and doxorubicin (VID), with G-CSF support, in children with newly diagnosed inoperable or metastatic non-rhabdomyosarcoma soft tissue sarcomas.

SECONDARY OUTCOMES:
Event-free Survival
  To estimate the 2-year survival and event-free survival of children treated with VID in combination with radiotherapy and/or surgery
Establish a bank of frozen tissue (tumor and peripheral blood)
  To establish a bank of frozen tissue (tumor and peripheral blood) for use in further molecular studies.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto S. Pappo, MD, Study Chair — St. Jude Children's Research Hospital
Locations (9):
- United States (7):
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland